CLINICAL TRIAL: NCT02879097
Title: Efficacy, Safety & Immunogenicity Study of CBT124 & EU-sourced Avastin® in Combination With Carboplatin and Paclitaxel in First-line Treatment in (NSCLC)
Brief Title: Efficacy-Safety-Immunogenicity Study of CBT124&EU-sourced Avastin® in Stage 4 NSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cipla BioTec Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBT124/CT/002; 2016-003301-34 (EudraCT Number)
Record Dates: First submitted 2016-08-16; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Non-Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT124 arm (Experimental): CBT124 plus carboplatin and paclitaxel
  Interventions: Biological: CBT124; Drug: Carboplatin; Drug: Paclitaxel
- EU Sourced Avastin® arm (Active Comparator): EU-sourced Avastin® plus carboplatin and paclitaxel
  Interventions: Biological: EU-sourced Avastin®; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Biological: CBT124 — Induction Phase: CBT124 15 mg/kg IV infusion-Day 1 of each 3-week Cycle for 6 cycles; Carboplatin AUC 6 mgXmin/mL (calculation-Calvert formula recommended) on Day 1 of each 3-week Cycle for 6 cycles; Paclitaxel 200 mg/m2 on Day 1 of each 3-week Cycle for 6 cycles. Maintenance Phase: All the subjects who complete the induction phase and are alive at Week 19 without progression of the disease can be included in the maintenance phase and receive CBT124 (bevacizumab, 15 mg/kg, intravenous infusion on Day 1 of each 3-week Cycle) up to disease progression or unacceptable toxicity (that precludes further treatment with bevacizumab) or death.
  Arms: CBT124 arm
Biological: EU-sourced Avastin® — Induction Phase: EU-sourced Avastin® 15 mg/kg IV infusion-Day 1 of each 3-week Cycle for 6 cycles; Carboplatin AUC 6 mgXmin/mL (calculation-Calvert formula recommended) on Day 1 of each 3-week Cycle for 6 cycles; Paclitaxel 200 mg/m2 on Day 1 of each 3-week Cycle for 6 cycles. Maintenance Phase: All the subjects who complete the induction phase and are alive at Week 19 without progression of the disease can be included in the maintenance phase and receive CBT124 (bevacizumab, 15 mg/kg, intravenous infusion on Day 1 of each 3-week Cycle) up to disease progression or unacceptable toxicity (that precludes further treatment with bevacizumab) or death.
  Arms: EU Sourced Avastin® arm
Drug: Carboplatin — Induction Phase: Carboplatin AUC 6 mgXmin/mL (calculation-Calvert formula recommended) on Day 1 of each 3-week Cycle for 6 cycles.
Drug: Paclitaxel — Induction Phase: Paclitaxel 200 mg/m2 on Day 1 of each 3-week Cycle for 6 cycles.

SUMMARY:
The purpose of this study is to determine whether CBT124 and Avastin® are comparable in terms of efficacy, safety, immunogenicity; and whether the pharmacokinetics of CBT124 matches that of Avastin® (pharmacokinetics is nested in this study for Indian patients).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether CBT124 and Avastin® are comparable in terms of efficacy, safety, immunogenicity; and whether the pharmacokinetics of CBT124 matches that of Avastin® (pharmacokinetics is nested in this study for Indian patients). To test the clinical equivalence in terms of efficacy and safety, a two-sided test approach based on a pre-specified range to test the null hypothesis that the proposed biosimilar is either (1) inferior to the reference product or (2) superior to the reference product based on the pre-specified equivalence margin will be used. The equivalence margins are chosen to enable detection of clinically meaningful differences in effectiveness between CBT124, candidate biosimilar bevacizumab and reference product (EU-sourced Avastin®) at the 95% confidence interval (CI). In this trial, asymmetric equivalence margins will be used, i.e., the upper (superiority) and the lower (inferiority) bounds of the equivalence margin are not symmetric. The goal is to reject the null hypothesis of non-equivalence and accept the alternative hypothesis that the two treatments (in this case, CBT124 and EU-sourced Avastin®) are equivalent (i.e., the differences between the two are not clinically and statistically meaningful). The hypothesis testing will be performed by determining if the difference in the primary end point (Objective Response Rate [ORR]) between the reference product (EUsourced Avastin®) and proposed biosimilar (CBT124) is within the equivalence margin at the 95% CI.

ELIGIBILITY:
Inclusion Criteria: Subjects may be entered in the study only if they meet all of the following criteria:

* Adult subjects aged ≥ 18 to 75 years (≥ 18 to 65 years for India) with histologically or cytologically confirmed advanced non-squamous NSCLC.
* Epidermal growth factor receptor (EGFR) negative or wild type mutations
* Stage IV (Unresectable recurrent disease or metastatic) NSCLC
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Evaluable disease status or measurable tumor
* Adequate hepatic, renal, and bone marrow function
* Subjects with pre-existing hypertension must be well controlled on a stable regimen of antihypertensive therapy. Have systolic blood pressure ≤ 140 and ≥ 90 mmHg, diastolic blood pressure ≤ 90 and ≥ 50 mmHg and heart rate ≥ 40 and ≤ 90 bpm at screening and admission.
* Ability to understand risks of participation in the study and willingness provide informed consent.

Exclusion Criteria: Subjects will not be entered in the study for any of the following reasons:

* Small cell lung cancer (SCLC) or combination of SCLC and NSCLC. Squamous-cell tumors and mixed adenosquamous carcinomas of predominantly squamous nature
* Prior therapy with monoclonal antibodies or small molecule inhibitors against VEGF or VEGF receptors, including bevacizumab
* Prior therapy with carboplatin or paclitaxel
* Prior systemic therapy for metastatic disease. Prior systemic anticancer therapy or radiotherapy for locally-advanced NSCLC if completed < 12 months prior to screening
* Evidence of a tumor that compresses or invades major blood vessels or tumor cavitation that in the opinion of the Investigator is likely to bleed
* Symptomatic brain metastasis
* Previous malignancy other than NSCLC in the last 5 years except for basal cell cancer of the skin or pre-invasive cancer of the cervix
* Any unresolved toxicity > Common Toxicity Criteria Grade 1 (except alopecia) from previous anticancer therapy (including radiotherapy)
* History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding. Thrombotic or hemorrhagic event ≤ 6 months prior to screening
* History of hemoptysis greater than ½ teaspoon of bright red (fresh) blood in the past 4 weeks
* Subjects receiving long-term aspirin (> 325 mg/day), or other non-steroidal anti-inflammatory agents, or other drugs known to inhibit platelet function, treatment with dipyridamole, ticlopidine, or clopidogrel
* Subjects receiving anticoagulants
* Subjects who plan to undergo surgery during the study period
* Subjects who have undergone a major surgery, or have had a significant traumatic injury within 4 weeks prior to randomization
* Subjects who have a significant non-healing wound, or bone fracture within 4 weeks prior to randomization
* Subjects with history of gastrointestinal perforation or fistula formation
* Subjects with known hypersensitivity to any of the ingredients of the investigational products, or mammalian cell-derived products
* Female subjects who are pregnant, breast-feeding, planning to be pregnant during the study, or women of child-bearing potential (any woman who is not surgically sterile i.e., bilateral tubal ligation, total hysterectomy or < 2 years post menopause) not using a reliable method of double contraception (e.g. condom plus diaphragm, condom or diaphragm plus spermicidal gel/foam, tubal ligation, or stable dose of hormonal contraception) throughout the study period
* Male subject with a partner of childbearing potential who does not consent to the use of a reliable method of double contraception
* Subjects with uncontrolled hypertension
* Subjects with active infection assessed to be clinically significant by Investigator
* Known history of, or positive test result for human immunodeficiency virus (HIV), hepatitis C virus (test for hepatitis C virus antibody [HCVAb]) or hepatitis B virus (test for Hepatitis B surface Antigen [HBsAg])
* History of alcohol or substance abuse
* Prior treatment with any investigational drug within the 30 days prior to screening, or within 5 half-lives of the drug, whichever is longer
* Inability to comply with study requirements
* Other unspecified reasons that, in the opinion of the Investigator or Sponsor, make the subject unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 19 weeks
  Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumours (RECIST) criteria (version 1.1). Defined as the proportion of subjects whose best confirmed overall response over Week 1 to Week 19 is either Complete Response (CR) or Partial Response (PR). Confirmed best overall response (complete or partial response) may be claimed only if the criteria for each are met after a repeat radiologic tumor assessment (using RECIST criteria version 1.1) 6 weeks later.

SECONDARY OUTCOMES:
Progression-free survival (PFS) rate at 1 year | 1 year
  Duration of response.
Overall Survival (OS) rate at 1 year | 1 year
  Duration of response.
Pharmacokinetics: Cmax and Ctrough | Cycle 6
  Cycle 1: Cmax; Cycle 2-6: Ctrough
Proportion of subjects with selected adverse events (AE) | 1 year
  Proportion of subjects with selected adverse events (AE) of gastrointestinal perforation, hypertension, proteinuria, and pulmonary haemorrhage
Proportion of subjects with other selected AEs | 1 year
  Proportion of subjects with other selected AEs of hemorrhages, wound healing complications, abscess, and fistula formation
Proportion of subjects with other selected AEs/ SAEs/ Vital signs/Lab abnormalities | 1 year
  proportion of subjects with other selected AEs of Anaphylactic/ hypersensitivity/ infusion-related reactions, arterial and venous thromboembolic events, and febrile neutropenia Incidence of AEs (overall), serious adverse events (SAEs), including changes in vital signs and laboratory abnormalities
Incidence of anti-drug (bevacizumab) antibody formation | 1 year
  Incidence of anti-drug (bevacizumab) antibody formation, including incidence of neutralizing antibodies; Analysis of anti-drug antibody (ADA) positive and negative sub-population for PK, safety and efficacy.
Analysis of anti-drug antibody (ADA) positive and negative sub-population for PK, safety and efficacy | 1 year
  Analysis of anti-drug antibody (ADA) positive and negative sub-population for PK, safety and efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Tamal Raha, PhD, Study Director — Cipla BioTec

IPD SHARING:
Plan to Share IPD: Undecided
Study CBT124/CT/002 does not have a FDA regulated intervention.